CLINICAL TRIAL: NCT06779110
Title: IN-Stent RestenosIs Detection and TrEtment by Optical Coherence Tomography
Brief Title: Intracoronary Optical Coherence Tomography Guidance Vs. Angiography Only Guidance for Treatment of Coronary In-stent Restenosis
Acronym: INSIDE OCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Luigi Gonzaga Hospital (Other)
Responsible Party: Principal Investigator, Enrico Cerrato, Principal Investigator, Medical Doctor, San Luigi Gonzaga Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 002-2023
Record Dates: First submitted 2023-04-27; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: Coronary Artery Disease; Stent Restenosis; STENT
Keywords: Percutaneous Coronary Intervention (PCI); Optimal Coherence Tomography (OCT)
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OCT arm (Group 1) (Active Comparator): PCI of ISR guided by OCT (group 1): in this case, the operator has to perform at least one OCT run before and one OCT run at the end of PCI. The operator is left free to review the OCT run in the console directly and is left free to perform during PCI any additional OCT run. Dedicated flow-chart of treatment should be followed by operator during PCI
  Interventions: Procedure: Percutaneous Coronary Intervention
- Angio arm (Group 2) (Active Comparator): PCI of ISR guided by angiography (group 2): in this case, the operator has to perform PCI following angiography. To allow outcome computation, OCT will also be performed in this group at the beginning and the end of PCI, although the operator will be wholly blinded to any OCT findings. A detailed description of the blinding modality is reported in the following paragraph.
  Interventions: Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — Using OCT to guide PCI in ISR

SUMMARY:
Although advances in drug-eluting stents (DES) have substantially reduced the risk of coronary in-stent restenosis (ISR) and the need for target lesion revascularisation (TLR), ISR persists. There are several treatment options for ISR (conventional balloon angioplasty, cutting or scoring balloons, drug-coated balloons, repeat DES implantation or bypass surgery). Coronary imaging is mandatory to perform PCI on ISR. Optimal coherence tomography (OCT) is an excellent option to guide PCI, but its role in ISR-PCI remains unclear. The INSIDE OCT Trial aims to compare the acute performance of PCI for ISR, either guided by OCT and angiography or by angiography alone.

DETAILED DESCRIPTION:
INSIDE-OCT is an investigator-initiated, randomised, multicenter, non-blinded trial.

Patients presenting with acute coronary syndrome or stable ischemic heart disease and ISR (angiographic stenosis between 70% and 99% in at least two projections, in a vessel with a lumen diameter ≥ 2.25 - ≤ 5.75 mm) with PCI indication will be randomised (1:1) to undergo either PCI guided by OCT (Group 1) or PCI with angiographic guidance only (Group 2).

Nowadays, PCI is performed following current guidelines and clinical practice. Any manoeuvre is left to the operator's discretion. Any approved intracoronary gears could be used (multiple wires, compliant, non-compliant, cutting, scoring balloons, Drug coated balloons, new stents implantation etc.).

Randomisation will be performed on the online eCRF site immediately after the end of the diagnostic angiography after acquiring the patient's study informed consent and after reviewing inclusion/exclusion criteria.

Randomisation will generate two groups:

PCI of ISR guided by OCT (group 1): in this case, the operator has to perform at least one OCT run before and one OCT run at the end of PCI. The operator is left free to review the OCT run in the console directly and is left free to perform during PCI any additional OCT run.

PCI of ISR guided by angiography (group 2): in this case, the operator has to perform PCI following angiography. To allow outcome computation, OCT will also be performed in this group at the beginning and the end of PCI. However, the operator will be wholly blinded to any OCT findings. A detailed description of the blinding modality is reported in the following paragraph.

Blinding: In Group 2, OCT will be performed at the beginning of the procedure, although the operator will be blinded to any OCT findings. In practice, the operator will perform OCT pullback properly, advancing the probe in the target vessel following angio guidance but without viewing the OCT monitor in the cath lab. A trained nurse/technician not involved in any decision regarding the procedure will guide the operator to perform an OCT pullback correctly and will check immediately if the OCT run is consistent with the current standard of quality. The operator could not receive any information from the OCT run recorded at this stage and had to proceed with the PCI procedure with angio-only guidance Therefore, the operator will declare the end of the procedure after completing all PCI manoeuvres judged necessary to obtain an excellent angiographic result. At this stage, an OCT pullback will be performed again to appraise OCT final data required for primary endpoint computation.

Therefore, the operator should evaluate the OCT runs, and he will be left free to perform additional PCI manoeuvres to optimise the result if necessary.

In groups 1 and 2, the operator should detail his PCI planned strategy before and after OCT runs. Changes in PCI planning after OCT disclosure will be recorded in both groups (see secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed
* Age ≥ 18 years
* Referred for angiography either in stable or ACS setting suitability for PCI through femoral or radial access
* A coronary in-stent restenosis between 70% and 99% in at least two projections in a vessel with a lumen diameter ≥ 2.25 - ≤ 5.75 mm (The severity of the stenosis should be based on visual estimation, with current online state-of-the-art angiographic equipment of the participating centres and after a mandatory dose of 50-200 mcg intracoronary of nitroglycerine.
* Stable hemodynamics

Exclusion Criteria:

* Inability to give informed consent
* Participation in another clinical study with an investigational product
* OCT pullback not technically feasible in vessel site

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Imaging Outcome (powered): Delta MSA defined as: cross Sectional Area (CSA,mm2) post-PCI minus CSA (mm2) at baseline in the same coronary restenotic segment, continuous measure | Periprocedural
  Delta MSA assessed by OCT (same frame) in each randomized arm, measured at an independent OCT core laboratory blinded to imaging modality assignment.

SECONDARY OUTCOMES:
Clinical outcome: MACE (Major Adverse Cardiovascular Events) in experimental vs control group | 1-year
  Time-to-first-event rate of the composite outcome of all cause of death, non-fatal MI, ID-TLR at 1 year in experimental group vs control group
Imaging Outcome: Delta MSA defined as: cross Sectional Area (CSA,mm2) post-PCI minus CSA (mm2) at baseline in the same coronary restenotic segment, continuous measure | Periprocedural
  Delta MSA assessed by OCT (same frame) in control (angio-guided) arm, in patients treated with additional manouvers after OCT disclosure, measured at an independent OCT core laboratory blinded to imaging modality assignment.
Number of cases in which additional PCI maneuvers was performed after disclosure of OCT pullback in the entire population | Periprocedural
  Additional PCI manouvers performed by operators after OCT disclosure including changings in size of balloons, any balloon dilatations, cutting/scoring, IVL, DEB, DES implantation
Number of intracoronary devices used in experimental vs control group (continuous, mean) | Periprocedural
  number of devices used including balloons stents and debulking devices
Quantitative flow ratio value (QFR, mean number) at the end of PCI in experimental vs control group, continuous | Periprocedural
  Mean Quantitative flow Ratio value assessed by QFR sofware in each randomized arm, measured at an independent core laboratory blinded to imaging modality assignment.

OTHER OUTCOMES:
Number of patient with device-related (OCT) complications in the whole population | periprocedural
  number of cases with perforations, dissections, abrupt vessel closure, TIMI flow reduction or other coronary complications related to advancement or retrieval or OCT probe pullback
Number of patient with acute kidney injury in the entire study population. | within hospitalization
  Acute kidney injury (AKI) was defined as the presence of any of the following (not graded): elevation in the serum creatinine level by >= 0.3 mg/dl within 48hours; or increase >= 1.5 times tnat at baseline or urine volume < 0.5 ml/kg/h for 6 hours
Clinical outcome: MACE (Major Adverse Cardiovascular Events) | within 1 year
  Time-to-first-event rate of the composite outcome of all cause of death, non-fatal MI, ID-TLR at 1 year in experimental group vs historical cohort of patients with ISR treated with angio-only guided PCI in the current DES generation

CONTACTS AND LOCATIONS:
Locations (12):
- Italy (12):
  - Osp Aosta, Aosta, Aosta
  - Biella, Biella, Biella
  - Osp. S. Croce e Carle, Cuneo, Cuneo
  - Ospedale Universitario di Ferrara, Cona, Ferrara
  - Osp Universitario S. Marino, Genova, Genova
  - Infermi Hospital, Rivoli ASLTO3, Rivoli, Italy
  - Ospedale di Trapani, Trapani, Trapani
  - AOU San Luigi Gonzaga, Orbassano, Turin
  - AO Mauriziano, Turin, Turin
  - AOU Città della Salute e della Scienza, Turin, Turin
  - Osp. Giovanni Bosco, Turin, TURIN
  - Osp Vercelli, Vercelli, Vercelli

IPD SHARING:
Plan to Share IPD: No